CLINICAL TRIAL: NCT06451354
Title: Postoperative Analgesia After Cesarean Section; Comparison Among Ultrasound Guided Erector Spinae, Quadratus Lumborum or Transversus Abdominis Plane Blocks: A Prospective Randomized Study
Brief Title: Postoperative Analgesia After Cesarean Section; Comparison Among Ultrasound Guided Erector Spinae, Quadratus Lumborum or Transversus Abdominis Plane Blocks
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Hasnaa Gamal Khafagy, Assistant Lecturer of Anesthesiology, Surgical Intensive Care and Pain Medicine, Faculty of Medicine, Kafrelsheikh University, Egypt., Kafrelsheikh University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 35439/4/22
Record Dates: First submitted 2024-06-02; First posted 2024-06-11 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Postoperative Analgesia; Cesarean Section; Erector Spinae Block; Quadratus Lumborum Block; Transversus Abdominis Plane Block
MeSH Terms: interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control group (No Intervention): Patients will receive the standard spinal anesthesia with 0.5% hyperbaric bupivacaine (2.2ml)
- Erector spinae plane block group (Experimental): Patients will receive bilateral ultrasound-guided erector spinae plane block after spinal anesthesia and at the end of surgery. The erector spinae plane block will be performed by using bupivacaine 0.25% (20 ml in each side). Erector spinae plane block will be performed at the level of T9.
  Interventions: Other: Erector spinae plane block (20 ml bupivacaine 0.25% in each side)
- Posterior Quadratus lumborum plane block group (Experimental): Patients will receive bilateral ultrasound-guided quadratus lumborum plane block after spinal anesthesia at the end of surgery. The quadratus lumborum plane block will be performed by using bupivacaine 0.25% (20 ml in each side).
  Interventions: Other: Posterior Quadratus lumborum plane block (20 ml bupivacaine 0.25% in each side)
- Lateral Transversus abdominis plane block group (Experimental): Patients will receive bilateral ultrasound-guided transversus abdominis plane block after spinal anesthesia at the end of surgery. The transversus abdominis plane block will be performed by using bupivacaine 0.25% (20 ml in each side) to the lateral abdominal wall in the mid-axillary line, between the lower costal margin and iliac crest.
  Interventions: Other: Lateral Transversus abdominis plane block (20 ml bupivacaine 0.25% in each side)

INTERVENTIONS:
Other: Erector spinae plane block (20 ml bupivacaine 0.25% in each side) — Patients will receive bilateral ultrasound-guided erector spinae plane block after spinal anesthesia and at the end of surgery. The erector spinae plane block will be performed by using bupivacaine 0.25% (20 ml in each side). Erector spinae plane block will be performed at the level of T9.
  Arms: Erector spinae plane block group
Other: Posterior Quadratus lumborum plane block (20 ml bupivacaine 0.25% in each side) — Patients will receive bilateral ultrasound-guided quadratus lumborum plane block after spinal anesthesia at the end of surgery. The quadratus lumborum plane block will be performed by using bupivacaine 0.25% (20 ml in each side).
  Arms: Posterior Quadratus lumborum plane block group
Other: Lateral Transversus abdominis plane block (20 ml bupivacaine 0.25% in each side) — Patients will receive bilateral ultrasound-guided transversus abdominis plane block after spinal anesthesia at the end of surgery. The transversus abdominis plane block will be performed by using bupivacaine 0.25% (20 ml in each side) to the lateral abdominal wall in the mid-axillary line, between the lower costal margin and iliac crest.
  Arms: Lateral Transversus abdominis plane block group

SUMMARY:
The aim of this prospective randomized controlled study is to compare the analgesic efficacy of the ultrasound-guided erector spinae plane block, ultrasound-guided quadratus lumborum plane block, and ultrasound-guided transversus abdominis plane block in patients undergoing elective cesarean section.

DETAILED DESCRIPTION:
Acute postpartum pain is a key determinant of maternal satisfaction; may lead to persistent postoperative pain.

Opioids are used to control severe pain. However, they have many common side effects as sedation, dizziness, nausea, vomiting, constipation, physical dependence, tolerance, and respiratory depression.

Transversus abdominis plane (TAP) block is a regional injection of local anesthetic between the transversus abdominis and internal oblique muscle planes. TAP block affects the sensory nerves of the anterolateral abdominal wall (T6-L1) that innervate the abdomen. TAP block is an easy technique, and decreases postoperative pain and opioid consumption.

Erector Spinae Plane block (ESPB), first described for analgesia in thoracic neuropathic pain has also been reported for the management of other causes of acute postoperative pain.

Quadratus Lumborum block (QLB) differ from the transversus abdominis plane block (TAP) it is a block of the posterior abdominal wall. It is also referred to as an inter fascial plane block because it requires the injection of a local anesthetic into the thoracolumbar fascia (TLF).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* American Society of Anesthesiologists (ASA) classification II.
* Female patients scheduled for elective cesarean section under spinal anesthesia.

Exclusion Criteria:

* Patient refusal.
* Patients who are taking analgesics for chronic illness or have history of substance abuse.
* Patients who are unable to describe their postoperative pain (e.g., language barrier or neuropsychiatric disorder).
* Patients with a history of coagulopathy.
* Patients weight less than 60 kilograms.
* Patient height less than 150 cm.
* Patients with known local anesthetics and opioid allergy.
* Patients with infection at the site of the needle puncture.
* Patients with major respiratory, cardiac, renal, or hepatic disorders.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Women undergoing elective cesarean section under spinal anesthesia.
Enrollment: 140 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
Postoperative morphine consumption | 24 hours postoperatively
  The rescue analgesia will be morphine IV bolus 3 mg with 5-minute lock out interval when Numeric Rating Scale (NRS)>3, can be repeated till NRS˂3 guided with the occurrence of complication.

SECONDARY OUTCOMES:
Degree of pain | 24 hours postoperatively
  Each patient will be instructed about postoperative pain assessment with the numeric rating scale (NRS) score. NRS (0 represents "no pain" while 10 represents "the worst pain imaginable"). NRS will be assessed at T1, 2, 4, 6, 12, 18, and 24 h postoperative.
Time for first request of the rescue analgesia | 24 hours postoperatively
  Time for first request of the rescue analgesia will be assessed from the end of surgery to first dose of morphine administrated.
Complications | 24 hours postoperatively
  Complications such as local anesthetic systemic toxicity (LAST), bradycardia, hypotension, nausea, vomiting, respiratory depression or any other complication will be recorded.
Degree of patient satisfaction | 24 hours postoperatively
  Degree of patient satisfaction will be assessed using 4-point scale (1, excellent; 2, good; 3, fair; 4, poor).

CONTACTS AND LOCATIONS:
Locations (1):
- Kafrelsheikh University, Kafr ash Shaykh, Kafrelsheikh, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.